CLINICAL TRIAL: NCT07039578
Title: An Open-Label, Multi-Center, Phase II Clinical Study Evaluating the Efficacy and Safety of CM336 Injection in the Treatment of Relapsed or Refractory Primary Light-Chain Amyloidosis
Brief Title: Study Evaluating the Efficacy and Safety of CM336 Injection in the Treatment of Light-Chain Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM336-026101
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Primary Light-Chain Amyloidosis
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose group(CM336) (Experimental)
  Interventions: Biological: CM336 Injection(Low dose group)
- High dose group(CM336) (Experimental)
  Interventions: Biological: CM336 Injection(High dose group)

INTERVENTIONS:
Biological: CM336 Injection(Low dose group) — subcutaneous CM336 administration, step-up dosing, Dose and frequency of CM336 according to the protocol.
  Arms: Low dose group(CM336)
Biological: CM336 Injection(High dose group) — subcutaneous CM336 administration, step-up dosing, Dose and frequency of CM336 according to the protocol.
  Arms: High dose group(CM336)

SUMMARY:
to Evaluate the Efficacy and Safety of CM336 (BCMA/CD3 Bispecific Antibody) in Adults with Relapsed or Refractory Primary Light-Chain Amyloidosis

ELIGIBILITY:
Inclusion Criteria:

* Voluntary provision of written informed consent and ability to comply with protocol requirements.
* Age ≥18 years, any gender.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
* Confirmed diagnosis of primary light-chain (AL) amyloidosis.
* Relapsed or refractory primary AL amyloidosis.
* Measurable hematologic disease at screening (per protocol-defined criteria).
* Involvement of ≥1 amyloid-affected organ.
* Adequate organ function meeting all protocol-specified criteria within 3 days prior to first dose.

Exclusion Criteria:

* Current or prior diagnosis of multiple myeloma.
* Received anti-AL amyloidosis therapy within protocol-specified timeframe prior to first dose.
* Clinically significant cardiovascular or cerebrovascular disease.
* Any active or uncontrolled infection meeting protocol-defined criteria.
* Any other condition deemed by the Investigator to preclude safe study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy after CM336 treatment | up to 3 years
  Hematologic complete response (hCR) rate

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Principal Investigator — Peking Union Medical College Hospital; Gang An, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality